CLINICAL TRIAL: NCT03740191
Title: "Spot-Scanning Based Hypofractionated Proton Therapy for Low and Intermediate Risk Prostate Cancer" "Hypofraktionierte Protonentherapie Mit Spot-Scanning-Technik Bei Prostatakarzinom Mit Niedrigem Oder Mittlerem Risiko"
Brief Title: Spot-Scanning Based Hypofractionated Proton Therapy for Low and Intermediate Risk Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recuitment target for patient enrollment was not met.
Sponsor: EBG MedAustron GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRLI-MA-012016; PRLI (Other: EBG MedAustron GmbH)
Record Dates: First submitted 2018-07-09; First posted 2018-11-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Low Risk Prostate Cancer; Intermediate Risk Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Therapy of Prostate Cancer (Other): Patients with low and intermediate risk are included. The following interventions are performed:
  * 'Expanded Prostate Cancer Index Composite' (EPIC) questionnaire
  * kV x-ray images
  * Conebeam CT
  Interventions: Other: EPIC questionnaire; Radiation: kV x-ray images; Radiation: Conebeam CT

INTERVENTIONS:
Other: EPIC questionnaire — The EPIC questionnaire is used to evaluated the Quality of life of the patients including the sexual function.
Radiation: kV x-ray images — After the applied daily fraction, x-ray imaging will be repeated daily to assess for intra-fraction motion of the prostate.
Radiation: Conebeam CT — For the assessment of interfraction target and organs at risk movement. Conebeam CT as soon as it becomes available will be performed 5 x/week or at each day of proton therapy before treatment application.

SUMMARY:
This prospective study assess the effectiveness and safety of hypofractionated proton radiotherapy in the treatment of intermediate and low risk prostate cancer.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness and safety of spot-scanning based hypofractionated proton radiotherapy for the treatment of intermediate and low risk prostate cancer. The treatment effectiveness is defined as freedom from biochemical failure. Treatment safety will be documented with acute and late morbidity assessments. Dose volume relationships for late side effects in organs at risk surrounding the prostate will be calculated from the dose volume histogram parameters assessed during treatment planning. Patient assessed Quality of life data including sexual function will be collected to increase our understanding how the reduction of normal tissue irradiation with proton therapy with subsequent decrease in functional impairments will overall affect the patient's life.

ELIGIBILITY:
Inclusion Criteria:

* Pathological (histologically) proven diagnosis of prostatic adenocarcinoma
* Clinical stage T1-T2b
* Prostate specific antigen (PSA) ≤ 20 ng/mL
* Gleason Score ≤ 7
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Clinically negative lymph nodes evaluated by imaging (pelvic +/- abdominal CT or MRI scan)
* Any patient with lymph nodes > 1.0 cm maximum diameter requires further studies to address eligibility. Positron emission tomography (PET)-CT is recommended for lymph nodes > 1.0 cm. Positive PET-CT indicates malignant involvement. Hence, the patient will be staged as "high-risk" and therefore declared ineligible for study participation. Negative PET-CT in lymph nodes 1.0-1,5 cm indicates non-involvement and thus eligibility. Negative PET-CT in lymph nodes > 1.5 cm is equivocal and requires additional work-up, preferably by biopsy.
* Patients must be 18 years of age or older. There is no upper age limit.
* Patient must be able to provide study-specific informed consent prior to study entry.
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) Questionnaire to assess Quality of Life.
* Previously initiated Androgen Deprivation Therapy (ADT) is acceptable.
* Patients with history of chronic bowel diseases may be included.
* Patients with previous Transurethral Resection of the Prostate (TURP) performed for urinary retention may be included.

Exclusion Criteria:

* Prior radiotherapy to the pelvic area.
* Prior prostate cancer therapy such as: prostatectomy, cryotherapy or hyperthermia.
* Prior systemic therapy (chemotherapy) for prostate cancer.
* Concurrent cytotoxic chemotherapy for prostate cancer.
* Evidence of distant metastases.
* Regional lymph node involvement.
* International Prostate Symptom Score (IPSS) > 20
* Hip prosthesis
* Second invasive malignancy (except of basal cell and squamous cell carcinoma of the skin in situ) if not controlled within last two years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
freedom from biochemical failure | 5 years
  Freedom from biochemical failure outcomes (FFBF) following spot-scanning based, moderately hypofractionated proton therapy will be compared with results of published studies using either similar or standard dose fractionation treatment regimen and using either photon or proton therapy. Determination of e.g., PSA, IPSS, Adverse Events

SECONDARY OUTCOMES:
Determination of the intra-fraction target movement using planar kilovoltage (kV) x-ray Imaging 5x/week or at each day of ion therapy. | daily through treatment completion (up to 4 weeks: from 1st day to last day of treatment)
Determination of the inter-fraction target and organ at risk movement using Conebeam CT 5x/week or at each day of ion therapy. | daily through treatment completion (up to 4 weeks: from 1st day to last day of treatment)
Determination of the incidence of gastrointestinal and genitourinary toxicities acute during treatment | weekly through treatment completion, Months 3(±1)
Determination of the incidence of gastrointestinal and genitourinary toxicities late at 2 years | Months 24(±2)
Determination of the incidence of gastrointestinal and genitourinary toxicities late at 5 years | Months 60(±4)
Assessment of the quality of life and sexual function following proton therapy. | Baseline, Months 3(±1), 6(±2), 12(±2), 18(±2), 24(±2), 36(±4), 48(±4), 60(±4)
  Change of quality of life and sexual function from Baseline following proton therapy. The Prostate cancer-specific Health-Related Quality of Life questionnaire Expanded Prostate Index Composite (EPIC-26) will be used. EPIC is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. EPIC-26 was developed as a short-form version of the full EPIC. This version contains 26 item and the same 5 domains as the full version of EPIC: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better quality of life.
Correlation of adverse events (toxicity), quality of life (QoL) and sexual function with dosevolume histogram parameters adjusted according to actual dose delivered. | Dose volume histogram parameters: Pre-Treatment, Toxicity: Weekly during proton therapy, Months 3(±1), 6(±2), 12(±2), 18(±2), 24(±2), 36(±4), 48(±4), 60(±4), Quality of life: Pre-Treatment, Months 3(±1), 6(±2), 12(±2), 18(±2), 24(±2), 36(±4)
  Correlation of adverse events (toxicity) (see Determination of the incidence of gastrointestinal and genitourinary toxicities), quality of life (QoL) and sexual function (see Assessment of the quality of life and sexual function) with dosevolume histogram parameters adjusted according to actual dose delivered.
Determine disease specific survival at 5 years. | 5 years
Determine overall survival at 5 years. | 5 years
Determination of the intra- and inter- mobility of prostate, seminal vesicles and rectum in order to further define and refine planning target volume parameters for future applications. | daily through treatment completion (up to 4 weeks: from 1st day to last day of treatment)
  Determination of the intra- and inter- mobility of prostate, seminal vesicles and rectum in order to further define and refine planning target volume parameters for future applications by using data assessed by determination of the intra-fraction target movement using planar kV x-ray imaging 5x/week or at each day of ion therapy (see Determination of the intra-fraction target movement using planar kilovoltage (kV) x-ray Imaging 5x/week or at each day of ion therapy) and determination of the inter-fraction target and organ at risk movement using Conebeam CT (see Determination of the inter-fraction target and organ at risk movement using Conebeam CT 5x/week or at each day of ion therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Carola Lütgendorf-Caucig, MD MPH MBA, Principal Investigator — EBG MedAustron GmbH
Locations (1):
- EBG MedAustron GmbH, Wiener Neustadt, Lower Austria, Austria